CLINICAL TRIAL: NCT00877994
Title: Breaking the Cycle of Risk: Intervention for Mothers With Eating Disorders
Brief Title: Nurture: A Program for Mothers With Histories of Disordered Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-0236; R34MH080750 (NIH)
Record Dates: First submitted 2009-04-06; First posted 2009-04-08 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Eating Disorders
Keywords: Disordered Eating; Parenting; Mothers
MeSH Terms: conditions — Feeding and Eating Disorders | interventions — Psychotherapy, Group

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate (Active Comparator): This group will receive the nurture group therapy immediately after enrolling in the study.
  Interventions: Behavioral: Nurture Support Group Therapy; Behavioral: Group therapy
- Delayed (Active Comparator): This group will receive the nurture group therapy 16 weeks after enrolling in the study.
  Interventions: Behavioral: Nurture Support Group Therapy; Behavioral: Group therapy

INTERVENTIONS:
Behavioral: Nurture Support Group Therapy — Participants will be randomly assigned (like the flip of a coin) to either receive the curriculum immediately (immediate group) or at a later time point approximately 16 weeks later (delayed group). Both groups will receive 16, 90 minute long group sessions delivered over 4 months. Groups will include 4-8 mothers and one or two co-therapists.
  Other Names: Parenting group
Behavioral: Group therapy — Participants will be randomly assigned (like the flip of a coin) to either receive the curriculum immediately (immediate group) or at a later time point approximately 16 weeks later (delayed group). Both groups will receive 16, 90 minute long group sessions delivered over 4 months. Groups will include 4-8 mothers and one or two co-therapists. The curriculum will focus on increasing positive healthy eating patterns in children of mothers who have had disordered eating and body image struggles.
  Other Names: Parenting groups

SUMMARY:
Nurture is a collaborative pilot study for mothers of children under the age of 3 who have suffered from disordered eating in the past. It is coordinated by the University of North Carolina at Chapel Hill, Duke University and Virginia Commonwealth University and sponsored by the National Institute of Mental Health. Nurture hopes to promote confident parenting and a positive meal times.

DETAILED DESCRIPTION:
Mothers who have struggled with disordered eating or body image struggles are often concerned how best to provide proper nutrition to their child and/or model healthy eating behavior. We have developed a curriculum that provides information about how to establish healthy eating patterns and social support for mothers with children under three years of age. The curriculum will be delivered in a support group format led by co-therapists affiliated with the UNC Eating Disorder Program.

ELIGIBILITY:
Inclusion Criteria:

* Has met lifetime DSM-IV criteria for anorexia nervosa (AN), bulimia nervosa (BN), or eating disorder not otherwise specified (EDNOS: including subthreshold AN, BN, and purging disorder, but excluding BED)
* BMI > 18.5 maintained for at least three months
* Has not met threshold criteria for AN or BN in the previous 28 days according to the Eating Disorders Examination, although subthreshold status or active residual symptomatology will not preclude entry
* Age 18 or older
* Has a child between the ages of 1 month and 2 years, 12 months old

Exclusion Criteria:

* Alcohol or drug dependence in the past year
* Current significant suicidal ideation reported during the assessment or on the BDI-II at baseline
* Developmental disability that would impair the ability of the participant to benefit from the intervention
* Psychosis, including schizophrenia, or bipolar I disorder
* Any families who have been the subject of social service inquiries

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Parenting self-efficacy | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Bulik, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Nancy Zucker, PhD, Principal Investigator — Duke University; Suzanne Mazzeo, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- University of North Carolina Chapel Hill, Chapel Hill, North Carolina, United States